CLINICAL TRIAL: NCT01740661
Title: Effects of Cryotherapy on Lower Extremity Joint Biomechanics During Running in Healthy Adults
Brief Title: Cryotherapy and Joint Biomechanics During Running
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Claudiane Fukuchi, BSc, PT, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IS-HPL-01
Record Dates: First submitted 2012-11-20; First posted 2012-12-04 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2013-01

CONDITIONS: Musculoskeletal Injury
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Cryotherapy (Experimental): The subjects will be exposed to a cold (~ 12° C) water immersion tub at the umbilical level for 20 minutes.
  Interventions: Other: Cryotherapy
- Control (Placebo Comparator): The subjects will be exposed to a non-cold (~ 26° C) water immersion tub at the umbilical level for 20 minutes.
  Interventions: Other: Control

INTERVENTIONS:
Other: Cryotherapy — The subjects will be exposed to a cold (~ 12° C) water immersion tub at the umbilical level for 20 minutes.
  Arms: Cryotherapy
Other: Control — The subjects will be exposed to a non-cold (~ 26° C) water immersion tub at the umbilical level for 20 minutes.
  Arms: Control

SUMMARY:
The purpose of this study is to determine the immediate effects of cryotherapy on the lower extremity biomechanics during running.

DETAILED DESCRIPTION:
Cryotherapy or cold therapy has widely been used as a treatment modality in both acute and chronic injuries. It is believe that the application of cryotherapy can help to decrease pain, muscle soreness, soft tissue swelling, and cause vasoconstriction of blood vessels reducing heat loss. The nerve conduction velocity and muscle-spindle firing rate also decreases with cryotherapy, which results in changes in proprioception acuity. Cryotherapy has also been used prior to exercise (pre-cooling) to improve endurance activities. However, given the possible detrimental effects of cryotherapy on proprioception acuity, the use of this treatment modality prior to exercise could pose an increased risk of musculoskeletal injury. The effects of cryotherapy on lower extremity biomechanics during athletic movements is poorly understood despite the wide use among physiotherapists, athletic therapists and clinicians. Therefore, the purpose of this investigation is to determine the effects of cold water immersion on lower extremity biomechanics during running. The investigators hypothesize that cryotherapy as a form of treatment can increase the load in the lower extremity joint during gait biomechanics.

ELIGIBILITY:
Inclusion Criteria:

* males or females (18 - 40 yrs)
* no injuries of the lower extremity in the past 6 months prior to participation
* recreationally active
* in good health upon entry into the study
* willing to volunteer for the present project.

Exclusion Criteria:

* lower extremity injury within the last 6 months
* circulatory, vestibular or any contradiction to cryotherapy including Raynaud's disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Knee frontal plane moments | 20 minutes
  Knee frontal plane loading will be calculated using inverse dynamics based on the ground reaction force data from a force plate and with kinematic data recorded by high speed cameras. Kinematics and kinetics data will be taken during running at 4m/s from each participant prior and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Performance Laboratory, University of Calgary, Calgary, Alberta, Canada